CLINICAL TRIAL: NCT02151630
Title: Comparison of 70% Pyruvic Acid Solution and Duofilm Solution in Treatment of Plantar Wart
Brief Title: Pyruvic Acid Versus Salicylic Acid Preparation in Treatment of Plantar Warts
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Fatima Assaf, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 393219
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Plantar Wart
Keywords: wart; verruca vulgaris; topical therapy; pyruvic acid; salicylic acid
MeSH Terms: conditions — Warts | interventions — Pyruvic Acid; Salicylic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pyruvic acid (Active Comparator): Patients will receive pyruvic acid solution 70% prepared by solving of pyruvic acid in water/ethanol solution. Patients will be advised to apply the solution twice daily for a period of four weeks. Application of petrolatum to the surrounding normal skin protects against the corrosive effect of the concentrated acid.
  Interventions: Drug: Pyruvic acid
- Salicylic acid (Active Comparator): Patients will receive a combination of salicylic acid 16.7%, lactic acid 16.7%, and collodion 100%. Patients will be advised to apply the solution twice daily for a period of four weeks. Application of petrolatum to the surrounding normal skin protects against the corrosive effect of the concentrated acid.
  Interventions: Drug: Salicylic Acid

INTERVENTIONS:
Drug: Pyruvic acid
  Arms: Pyruvic acid
Drug: Salicylic Acid
  Arms: Salicylic acid

SUMMARY:
Plantar warts can be bothersome and painful requiring treatment. The investigators will compare the efficacy of pyruvic acid and salicylic acid in treating multiple plantar warts. Patients with multiple plantar warts will be randomized to receive either pyruvic acid 70% or compound salicylic acid solution (salicylic acid 16.7%, lactic acid 16.7%, and collodion 100%) applying topically twice a day for 4 weeks. Patients will be visited every 2 weeks for one month after starting treatment and then every one month for up to 3 months. The number and size of warts will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* aged 12 years and above
* multiple warts (at least 2)

Exclusion Criteria:

* mosaic warts
* already under any treatment for warts
* pregnant or lactating women

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Wart number | From before to 3 months after
  Patients will be visited every two weeks for one month and then every month for up to 3 months by a dermatologist. On each visit, warts will be inspected to determine the number of warts. Any wart totally non-detectable by inspection and touch will be considered as healed.
Wart size | From before to 3 months after
  Patients will be visited every two weeks for one month and then every month for up to 3 months by a dermatologist. On each visit, warts will be inspected to determine the size of warts. The size of the warts will be calculated as the mean size of all the warts.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Assaf, M.D., Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Skin Diseases and Leishmaniasis Research Center, Isfahan, Isfahan, Iran

REFERENCES:
- [Background] Kwok CS, Holland R, Gibbs S. Efficacy of topical treatments for cutaneous warts: a meta-analysis and pooled analysis of randomized controlled trials. Br J Dermatol. 2011 Aug;165(2):233-46. doi: 10.1111/j.1365-2133.2011.10218.x. Epub 2011 May 26. PMID 21219294